CLINICAL TRIAL: NCT03221023
Title: Intrawound Vancomycin Prophylaxis During Stimulator Re-Implantation: A Multi-Center Randomized Controlled Trial
Brief Title: Intrawound Vancomycin Prophylaxis for Neural Stimulator
Acronym: IV-DIRT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Honey, Neurosurgeon, Professor of Surgery (Neurosurgery), Director of Surgical Centre for Movement Disorders, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H16-01496
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Vancomycin; Implantable Neural Stimulator; Deep Brain Stimulation; Surgical Site Infection
Keywords: Vancomycin; Implantable Neural Stimulator; Deep Brain Stimulation; Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Vancomycin; Saline Solution

STUDY DESIGN:
Intervention Model Description: The subjects meeting the inclusion criteria will be randomized to either the treatment arm or the control arm by site in a 1:1 ratio.
Who Masked: Participant, Care Provider
Masking Description: Both patient and surgeon will be blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vancomycin (Experimental): These patients will receive intrawound Vancomycin-saline and IV antibiotics
  Interventions: Drug: Vancomycin Hydrochloride; Drug: Saline Solution
- Saline (Placebo Comparator): These patients will receive intrawound saline + IV antibiotics alone
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Vancomycin Hydrochloride — Individuals in the experimental arm will receive intrawound Vancomycin-saline + IV antibiotics
  Arms: Vancomycin
Drug: Saline Solution — Individuals in the control arm will receive intrawound saline solution

SUMMARY:
The implantable pulse generator (IPG) is a device that generates electrical current to stimulate the spine, heart, or brain for various chronic conditions. In neurosurgery, the IPG is implanted in a subcutaneous pocket under the collarbone. This pocket is highly avascular and thus, antibiotics administered intravenously cannot reach a potential surgical site infection (SSI). SSIs cause millions of health care dollars to be wasted due to repeat surgery and hospital re-admissions. The investigators hope to to determine the effects of "intrawound vancomycin-saline and IV antibiotics" compared to "saline and IV antibiotics" on the incidence of IPG SSI rates 6-months post-surgery.

DETAILED DESCRIPTION:
Patients requiring neurosurgical IPG replacements will be recruited into this trial on a volunteer basis. The participants meeting the inclusion criteria will be randomized to either the treatment arm (intrawound Vancomycin-saline + IV antibiotics) or control arm (intrawound saline + IV antibiotics alone) by site in a 1:1 ratio. A sample size calculation using STplan determined that 405 patients per arm is required to reduce overall infection rate from 3.5% to 0.5% (80% power, α=0.05, two-tailed). Final sample size per arm will be 410 after generously accounting for loss to follow-up, non-compliance, and unrelated death.

The primary outcome will be a binary Yes/No on if IPG explantation due to infection was required within 6-months post-surgery.

This is a superiority trial and the investigators hypothesize intrawound Vancomycin-saline + IV antibiotics is superior to intrawound saline + IV antibiotics alone. An intention-to-treat analysis will be applied in a blinded manner once all patients have completed the trial and the database is locked.

The results of this trial will not only be applicable to neurosurgery, but also spine and cardiology.

ELIGIBILITY:
Inclusion Criteria:

* individuals who require INS replacement from Dr. C.R. Honey
* individuals who are between the ages of 18 to 80.
* individuals who consent to report any redness or swelling to their primary caregiver and follow-up as requested by their surgeon
* individuals who consent to keeping the study team informed of any medical concerns they may have regarding their INS for a minimum of 6 months postoperatively
* individuals who are capable of providing informed consent

Exclusion Criteria:

* individuals who have a history of autoimmune disease
* individuals who are undergoing any surgery or procedural intervention within six-months post-operatively of entrance into this study
* individuals who are on immunosuppression or any medication that would influence infection susceptibility
* individuals who are allergic to Vancomycin or Cefazolin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Device explantation 6 months post surgery | 6 months
  The primary outcome measure will be determined at the 6 month post surgery point, where the binary yes/no question, "was the INS device explanted", will be answered.

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doshi PK. Long-term surgical and hardware-related complications of deep brain stimulation. Stereotact Funct Neurosurg. 2011;89(2):89-95. doi: 10.1159/000323372. Epub 2011 Feb 2. PMID 21293168
- [Background] Caroom C, Tullar JM, Benton EG Jr, Jones JR, Chaput CD. Intrawound vancomycin powder reduces surgical site infections in posterior cervical fusion. Spine (Phila Pa 1976). 2013 Jun 15;38(14):1183-7. doi: 10.1097/BRS.0b013e31828fcfb5. PMID 23474597
- [Background] Martin JR, Adogwa O, Brown CR, Kuchibhatla M, Bagley CA, Lad SP, Gottfried ON. Experience with intrawound vancomycin powder for posterior cervical fusion surgery. J Neurosurg Spine. 2015 Jan;22(1):26-33. doi: 10.3171/2014.9.SPINE13826. PMID 25380539
- [Background] Ghobrial GM, Cadotte DW, Williams K Jr, Fehlings MG, Harrop JS. Complications from the use of intrawound vancomycin in lumbar spinal surgery: a systematic review. Neurosurg Focus. 2015 Oct;39(4):E11. doi: 10.3171/2015.7.FOCUS15258. PMID 26424335